CLINICAL TRIAL: NCT00114283
Title: A Phase 2 Trial of GW572016 in Patients With Metastatic and Recurrent Squamous Cell Carcinomas of the Head and Neck
Brief Title: Lapatinib Ditosylate in Treating Patients With Metastatic or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03823; NCI-2011-03823 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEAD AND NECK 04-3; UVACC-33604; CDR0000430924; NCI-6697; UVACC-HIC-11569 (Other: University of Virginia); 6697 (Other: CTEP); R21CA114986 (Other: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2012-11

CONDITIONS: Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive lapatinib ditosylate PO QD. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well lapatinib ditosylate works in treating patients with metastatic or recurrent head and neck cancer. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to estimate the objective response rate (complete response [CR] + partial response [PR]) in patients with squamous cell carcinomas of the head and neck following treatment with GW572016 (lapatinib ditosylate).

SECONDARY OBJECTIVES:

I. Secondary objectives of this study are to estimate time to progression, describe the adverse event profile, and to obtain preliminary assessments of changes in pre- versus post-treatment measurements for selected biomarkers in tumor cells from these patients.

OUTLINE:

Patients receive lapatinib ditosylate orally (PO) once daily (QD). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or recurrent squamous cell carcinoma of the head/neck; these include tumors arising in the oral cavity, oropharynx, nasopharynx, hypopharynx, glottis, or ethmoid/maxillary sinus; patients with localized disease must have failed primary therapy radiotherapy, surgery, and/or chemotherapy); patients with single site or regional recurrence that, in view of the Principal Investigator (PI) or treating physician is potentially curable by resection or by re-irradiation program, must have declined such therapies
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan; one or more sites of metastatic or recurrent disease must be accessible for needle biopsy
* No more than 2 prior chemotherapy regimens; no prior treatment with tyrosine kinase inhibitors or antibodies to the epidermal growth factor receptor (EGOR) or human epidermal growth factor receptor 2 (HER2)/neu; prior chemotherapy or radiation therapy completed at least 4 weeks prior to treatment with GW572016
* Life expectancy of greater than three months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes > 3,000/uL
* Absolute neutrophil count > 1,500/uL
* Platelets > 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or multigated acquisition (MUGA) scan; note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution
* Eligibility of patients receiving medications or substances known to affect, or with the potential to affect the activity or pharmacokinetics of GW572016 will be determined following review of their use by the Principal Investigator; patients requiring oral anticoagulants (coumadin, warfarin) are eligible provided there is increased vigilance with respect to monitoring international normalized ratio (INR); if medically appropriate and treatment available, the investigator may also consider switching these patients to low molecular weight (LMW) heparin, where an interaction with GW572016 is not expected
* The effects of GW572016 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Able to retain and absorb medication given by mouth or feeding tube

Exclusion Criteria:

* Prior treatment:

  * Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or
  * Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
  * Patients who have had prior treatment with EGFR targeting therapies
* Patients may not be receiving any other investigational agents or receiving concurrent anticancer therapy
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because GW572016 is member of the 4-anilinoquinazoline class of kinase inhibitors with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with GW572016, breastfeeding should be discontinued if the mother is treated with GW572016; human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with GW572016; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients with gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Concomitant requirement for medication classified as cytochrome P450 3A4 (CYP3A4) inducer or inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of antitumor activity as measured by objective response (CR+PR) evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) | At least 6 months
  Response will be classified by type and duration and 95% confidence intervals, adjusted for the interim looks, will be calculated.

SECONDARY OUTCOMES:
Adverse events will be classified by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 | Up to 12 months
  At study closure, adverse events will be classified by type, grade, duration and probable relation to treatment.
Time to progression evaluated using the RECIST | Time from start of treatment until disease progression or date of last follow-up, up to 12 months
  Product limit method will be used to estimate time to progression. We will have approximately 84% power to test the alternative with a one-sided 5% level test.
Changes in biochemical response as measured by biomarker data | Up to 12 months
  A proportional hazard model will be used to determine the association of selected markers with time to progression.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Thomas, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States